CLINICAL TRIAL: NCT04187274
Title: Evaluation of the Urethral Photoplethysmography-derived Perfusion Device (IKORUS) in Patients Undergoing Major Abdominal Surgery
Brief Title: Evaluation of the IKORUS Technology in Patients Undergoing Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Other Study IDs: P2019323
Record Dates: First submitted 2019-12-01; First posted 2019-12-05 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IKORUS technology — Ikorus technology is a new micro perfusion device measuring via urethral photoplethysmography, the urethral perfusion index (uPI) in patients equipped with an urinary catheter.

SUMMARY:
The goal of this observational substudy is to evaluate the feasibility, performance and behavior of the IKORUS (Advanced Perfusion Diagnostics, Villeurbanne, France), a new tissue perfusion device using urethral photoplethysmography in patients undergoing major abdominal surgery and in whom an advanced hemodynamic monitoring is placed.

DETAILED DESCRIPTION:
Continuous monitoring of tissue perfusion in patients undergoing major surgery remains challenging because of the lack of tools available. Through using urethral photoplethysmography, the urethral perfusion index (uPI) could allow tissue perfusion monitoring through a modified urinary catheter. The goal of this observational study is to evaluate the feasibility , performance and behavior of the IKORUS (Advanced Perfusion Diagnostics, Villeurbanne, France), a new device in the field. We aimed to assess its performance (duration and signal quality), the uPI variations during hemodynamic events (fluid challenge) in patients undergoing major abdominal surgery and equipped with an advanced hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing major abdominal surgeries and equipped with an advanced hemodynamic monitoring for goal directed therapy

Exclusion Criteria:

* Atrial fibrillation
* Ejection fraction < 30%

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Analysis of uPi evolution during surgery and comparison with Stroke volume | during surgery
  Percentage of case time with positive correlation between both variables (positive or negative) during a fluid challenge and during the whole case

SECONDARY OUTCOMES:
Occurrence of decreased perfusion during surgery | during surgery
  Occurrence of decreased perfusion during surgery

CONTACTS AND LOCATIONS:
Overall Officials: JOOSTEN ALEXANDRE, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme Hospital, Brussels, Brussel-hoofdstad, Belgium

IPD SHARING:
Plan to Share IPD: No